CLINICAL TRIAL: NCT04121026
Title: Validation of a Tuberculosis Treatment Decision Algorithm in HIV-infected Children
Brief Title: Validation of a Tuberculosis Treatment Decision Algorithm in HIV-infected Children (TB-Speed HIV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C18-27
Record Dates: First submitted 2019-10-01; First posted 2019-10-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis; HIV
Keywords: Tuberculosis; Diagnosis; HIV; Child
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Intervention Model Description: TB-Speed HIV is a prospective, multicentre management study evaluating the safety and feasibility of the recently proposed PAANTHER TB treatment decision algorithm for HIV-infected children with presumptive TB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: External validation of the PAANTHER TB treatment decision algorithm — The PAANTHER algorithm will be used for a TB treatment decision by site clinicians in all children enrolled in the study. The PAANTHER algorithm and prediction score was designed as a guiding tool for empirical TB treatment decision in HIV-infected children with presumptive TB. The proposed score includes:
  * history of contact
  * suggestive TB symptoms
  * tachycardia
  * chest radiography
  * abdominal ultrasound
  * Xpert MTB/RIF Ultra.
  A score of >100 is highly predictive of TB. In children with a score >100, anti-TB treatment will be initiated immediately. In children with a score of <100, TB treatment will not be initiated except in those with severe/life-threatening conditions for whom TB treatment decision could be made at the discretion of the site clinician. TB could be definitely ruled out after further assessment and decision made as to what treatment the children should receive in accordance with existing national protocols, along with clinical follow-up.

SUMMARY:
TB-Speed HIV is a prospective multicentre management study evaluating the safety and feasibility of the recently proposed PAANTHER TB treatment decision algorithm for HIV-infected children with presumptive TB. It will be conducted in four countries with high and very high TB (Tuberculosis) incidence (Côte d'Ivoire, Uganda, Mozambique, and Zambia) which have not participated in the study that developed the PAANTHER algorithm.

DETAILED DESCRIPTION:
The ANRS 12229 PAANTHER 01 (Pediatric Asian African Network for Tuberculosis and HIV Research) study, which enrolled 438 HIV-infected children of median age 7.3 (IQR: 3.3 - 9.7) years with presumptive TB in four countries (Burkina Faso, Cameroon, Cambodia, Vietnam) from 2011 to 2014, aimed at developing a diagnostic prediction score and algorithm for TB treatment decision in HIV-infected children. This was the first study developing a TB diagnostic score exclusively in HIV-infected children, using methods recommended for diagnostic prediction models. Based on microbiological, clinical and radiological features, the best scoring system obtained had a sensitivity of 88.6% and specificity of 61.2% when Xpert MTB/RIF was included in the algorithm. The investigators showed previously that mortality is high in children with both confirmed and unconfirmed TB and that initiation of anti-TB treatment, that occurred at a median time of 7 (IQR: 5 - 11) days in the study, led to delayed ART initiation, which is associated to significantly increased mortality. The score, based on easily collected clinical features, chest radiographic features, Xpert MTB/RIF results, and abdominal ultrasonography, could enable same-day TB treatment decision. Abdominal ultrasonography has shown promise for the diagnosis of TB in both HIV-infected adults and children. In the PAANTHER study, it detected abdominal lymphadenopathy in 50% of culture confirmed TB cases and 35% of all confirmed and unconfirmed cases, with a specificity of 85%.

Developed in tertiary research-experienced health facilities, the PAANTHER score could enable standardized treatment decision in HIV-infected children with presumptive TB, and could be recommended for extensive use in secondary and primary healthcare settings where most of these children are seeking care. However, external validation studies are now needed to assess the predictive performance of the PAANTHER diagnostic score on independent datasets.

The PAANTHER TB treatment decision algorithm will be used for a TB treatment decision by site clinicians in all children enrolled in the study. Validation of the algorithm will be performed by evaluating the safety of withholding TB treatment in children not initiated on treatment as per the PAANTHER TB treatment decision algorithm. The safety of this strategy will be carefully assessed through review of safety reports every 4 to 6 months during study conduct by the safety sub-committee of the SAB.

Occurrence of algorithm failures in terms of missed TB cases (TB cases subsequently detected among untreated cases, i.e. false negatives) and cases with unlikely TB among those initiated on TB treatment as per the algorithm (cases not secondarily validated as confirmed or unconfirmed TB cases by the expert committee, i.e. false positives) will enable to estimate the negative and positive predictive values of the algorithm.

A centralized international Expert Committee will clinically review and validate TB diagnosis in children. This will enable assessment of the added value of new markers (MLR and CRP) and, if need be, to propose a new version of the score based on an optimised predicted probability.

The TB-Speed HIV study will be implemented in 7 tertiary healthcare level hospitals in capital cities of Côte d'Ivoire, Uganda, Mozambique, and Zambia. A total of 550 HIV-infected children (aged < 15 years) with clinically suspected TB (presumptive TB) will be enrolled, using standard entry criteria. The inclusion period will last until all sites have reached the expected number of children enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 month to 14 years
2. Documented HIV-infection (i.e., confirmed before entry into the study)
3. Presumptive TB based on at least one criteria among the following:

   1. Persistent cough for more than 2 weeks
   2. Persistent fever for more than 2 weeks
   3. Recent failure to thrive (documented clear deviation from a previous growth trajectory in the last 3 months or Z score weight/age < 2)
   4. Failure of broad spectrum antibiotics for treatment of pneumonia
   5. Suggestive CXR features

   OR

   History of contact with a TB case and any of the symptoms listed under point 3 with a shorter duration (< 2 weeks)
4. Informed consent signed by parent/guardian

Exclusion Criteria:

Ongoing TB treatment or history of intake of anti-TB drugs in the last 3 months (isoniazid alone or rifampin/isoniazid for preventive therapy is not an exclusion criteria)

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Proportion of missed TB cases | 6 months
  Proportion of missed TB cases (false negative cases) in children not initiated on treatment as per the PAANTHER TB treatment decision algorithm

SECONDARY OUTCOMES:
Feasibility of the PAANTHER TB treatment decision algorithm (a): Proportion of children with presumptive TB having completed the algorithm. | 6 months
  The algorithm will be considered completed if a decision to initiate TB treatment has been taken at any step of the algorithm or if TB has been excluded after systematic evaluation, and all steps planned in the algorithm have been implemented.
Feasibility of the PAANTHER TB treatment decision algorithm (b): Time to final TB treatment decision | 6 months
Proportion of HIV-infected children with unlikely TB among those initiated on treatment as per the PAANTHER TB treatment decision algorithm | 6 months
  Proportion of cases considered as unlikely TB by the Expert Committee in those initiated on treatment as per the PAANTHER TB treatment decision algorithm (false positive)
Incidence of morbidity | 6 months
  Incidence of morbidity defined as drug-induced toxicity (ART and TB treatment-related), opportunistic infections, and IRIS, with or without TB treatment
Incidence of mortality | 6 months
Time to ART initiation in ART-naïve children | 6 months
CD4 (absolute count and %) gain | 6 months
  Immunologic evolution at 6 months after enrolment defined as CD4 cells gain (absolute count and %)
TB treatment outcomes (a): Weight gain at 6 months (absolute value and percentage of body weight) | 6 months
  TB treatment outcome in HIV-infected children initiated on treatment as per the PAANTHER TB treatment decision algorithm defined by weight gain at 6 months (absolute value and percentage of body weight)
TB treatment outcomes (b): TB symptoms resolution in children on TB treatment | 6 months
Feasibility of IPT initiation (a): Time to IPT initiation | 6 months
  Time to Isoniazid Preventive Therapy (IPT) initiation in HIV-infected children not initiated on treatment as per the PAANTHER TB treatment decision algorithm (a)
Feasibility of IPT initiation (b): Proportion of children initiated on IPT | 6 months
  Proportion of children initiated on IPT in HIV-infected children not initiated on treatment as per the PAANTHER TB treatment decision algorithm (b)
Performance of the Monocyte-to-Lymphocyte Ratio and the C-reactive protein and their potential added value in the PAANTHER score and algorithm to detect TB | 6 months
  Discrimination (area under the receiver-operating-characteristic curves [AUROC]) and calibration measures of the PAANTHER prediction model including or not MLR and CRP, against the TB composite reference standard as defined by the Expert Committee
Proportion of NPAs (or sputum) and stool samples with mycobacterium tuberculosis (MTB) detected using Ultra | 6 months
  Diagnostic performance of Ultra performed on one NPA and one stool sample against mycobacterial culture performed on standard samples in HIV-infected children
Proportion of children with NPA and stool samples collected as per study protocol | 6 months
  Feasibility of NPA and stool samples collection in HIV-infected children defined as the proportion of children with NPA and stool samples collected as per study protocol
Proportion of NPA-related adverse events (AEs) | 6 months
  Safety of NPA collection defined as proportion of AEs (vomiting, nose bleeding, low oxygen saturation, respiratory distress) occurring during NPA
Discomfort/pain/distress experienced by the child during NPA as assessed by the child | Within 3 days of inclusion
  Tolerability of NPA collection defined as discomfort/pain/distress experienced by the child during NPA, as assessed by the child using the Wong-Baker face scale (in a subset of children).
  Scale range: 0 (no hurt) - 5 (hurts worst)
Discomfort/pain/distress experienced by the child during NPA as assessed by the parents | Within 3 days of inclusion
  Tolerability of NPA collection defined as discomfort/pain/distress experienced by the child during NPA, as assessed by the parents using the visual analog scale (in a subset of children).
  Scale range: 0 (no pain) - 10 (pain as bad as it could possibly be)
Discomfort/pain/distress experienced by the child during NPA as assessed by the nurse | Within 3 days of inclusion
  Tolerability of NPA collection defined as discomfort/pain/distress experienced by the child during NPA, as assessed by the nurses using the "Face Legs Activity Cry Consolability" behavioral pain scale (in a subset of children).
  Total score range: 0 (relaxed and comfortable) - 10 (severe discomfort/pain). Each item of the FLACC scale - Face, Legs, Activity, Cry, Consolability - has 3 possible quotes: 0 or 1 or 2, with a precise description provided to help with the rating. The total score is obtained by adding individual item scores.
Sensitivity | 6 months
  false negative rate, i.e. negative predictive value, and corresponding sensitivity of the PAANTHER algorithm in the different subgroups in terms of age, CD4 counts, nutritional statuses, and timings of ART initiation (on/off ART)
Positivity | 6 months
  false positiverate, i.e. Positive predictive value, and corresponding positivity of the PAANTHER algorithm in the different subgroups in terms of age, CD4 counts, nutritional statuses, and timings of ART initiation (on/off ART)

OTHER OUTCOMES:
Incremental cost-effectiveness ratio (ICER) | 33 months
  Incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marcy, MD, PhD, Principal Investigator — University of Bordeaux, France; Maryline Bonnet, MD, PhD, Principal Investigator — Institut de Recherche pour le Développemnt (IRD) Montpellier, France; Eric Wobudeya, MD, PhD, Principal Investigator — MU-JHU Care Ltd, Kampala, Uganda
Locations (7):
- Côte d’Ivoire (2):
  - Cocody University Teaching Hospital, Abidjan
  - Treichville University Teaching Hospital, Abidjan
- Mozambique (2):
  - José Macamo General Hospital, Maputo
  - Maputo Central Hospital, Maputo
- Mbarara Regional Hospital, Mbarara, Uganda
- Zambia (2):
  - Lusaka University Teaching Hospital, Lusaka
  - Arthur Davidson Children Hospital, Ndola

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: TB-Speed project official website — https://www.tb-speed.com